CLINICAL TRIAL: NCT01721538
Title: Secondary Prevention of Stroke Through Participation in the Non-drug Therapeutic Weight Reduction Program: A Single-blinded Randomized Controlled Multicenter Trial
Brief Title: Secondary Prevention of Stroke Through Non-drug Therapeutic Weight Reduction
Acronym: SCENARIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Collaborators: Von Behring-Röntgen Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Yaroslav Winter, Neurologist and Research Fellow, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCENARIO OP1
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Stroke; Obesity
Keywords: stroke; prevention; obesity; weight reduction
MeSH Terms: conditions — Stroke; Obesity; Weight Loss | interventions — Weight Reduction Programs

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapy arm (Experimental): Non-drug therapeutic weight reduction program (15 weeks)
  Interventions: Other: Weight reduction program
- Control arm (Placebo Comparator): Lecture on healthy nutrition (1 hour)
  Interventions: Other: Lecture on healthy nutrition

INTERVENTIONS:
Other: Weight reduction program
  Arms: Therapy arm
Other: Lecture on healthy nutrition
  Arms: Control arm

SUMMARY:
SCENARIO is a trial to investigate the role of non-drug weight reduction in secondary prevention of stroke. It is a single-blinded, randomized, controlled multicentre trial with two arms. The therapy arm is participating in a comprehensive weight reducing program, whereas the control group takes part in a lecture on healthy nutrition. The primary study objective is to assess the efficacy of non-drug therapeutic weight reduction in the secondary prevention of stroke. Secondary objectives are functional outcome, cognitive status, post stroke depression, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke
* Age: 20 - 85 years
* BMI ≥ 25.0 kg/m² or waist circumference in men ≥ 94cm and in women ≥ 80cm
* Functional impairment, which would allow to participate in weight reduction program (mRS 0-4, NIHSS 0-12)
* Patient must be capable of understanding informed consent
* Written informed consent for participation in the study

Exclusion Criteria:

* Intracerebral hemorrhage as primary cause of stroke (secondary hemorrhage is not an exclusion criterion)
* Speech disturbance (aphasia or sever dysarthria)
* Dimming of consciousness
* Stroke due to arterial dissection or coagulation disorder
* Drug-related weight changes during previous 3 months
* Changes in appetite influencing medication listed in appendix during previous 3 months
* Bariatric surgery in the past
* Diabetes mellitus with a history of severe ketoacidosis
* Pregnancy or nursing
* Severe co-morbid disorders, e.g.:

  * AV-Block ≥ 2nd degree
  * Heart insufficiency (NYHA > 2)
  * Pericarditis, pericardial effusion
  * Severe kidney insufficiency (Creatinine > 3 mg/dl; Urea > 150 mg/dl)
  * Hepatic insufficiency (GOT > 3 x ULN; GPT > 3 x ULN)
  * Severe psychiatric disease within the last six months (psychosis, suicide attempts)
  * Chronic alcohol addiction or drug addiction
  * HIV- or hepatitis infection
  * Bleeding peptic ulcer (unless there is radiological evidence of healing 6 months prior to start of obesity program)
* Cognitive impairment with MMSE < 20
* Depression with BDI > 20
* Patients who are unable to give consent to study participation (MMSE < 20, aphasia)
* Recurrent stroke or myocardial infarction in the period between screening for study participation and start of weight reduction program
* Simultaneous participation in another clinical trial

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the number of deaths or major vascular events defined as stroke, TIA, myocardial infarction or hospitalization due to angina pectoris, which occur between the randomization and last follow-up. | 18 months

SECONDARY OUTCOMES:
Functional outcome | 18 months
  Functional outcome as measured by the modified Rankin Scale (mRS), NIH Stroke Scale (NIHSS) and Barthel Index (BI)
Cognitive deficits | 18 months
  Cognitive deficits in terms of vascular dementia as measured by the Structural Interview for diagnosis of Alzheimer dementia and multi-infarct dementia (SIDAM), the Vascular Dementia Assessment Scale cognitive subscale (VADAS-Cog), Stroop test and the Trail Makin Test
Post stroke depression | 18 months
  Post stroke depression as measured by Beck Depression Inventar (BDI II) and health-related quality of life (HrQoL) as measured by the EuroQol (EQ5D, visual analogue scale), Stroke Specific Quality of Life Scale, Stroke Impact Scale.
Severity of arterial hypertension, diabetes mellitus and hyperlipidemia | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Philipps-University Marburg, Marburg, Germany

REFERENCES:
- [Background] Winter Y, Rohrmann S, Linseisen J, Lanczik O, Ringleb PA, Hebebrand J, Back T. Contribution of obesity and abdominal fat mass to risk of stroke and transient ischemic attacks. Stroke. 2008 Dec;39(12):3145-51. doi: 10.1161/STROKEAHA.108.523001. Epub 2008 Aug 14. PMID 18703800